CLINICAL TRIAL: NCT02768272
Title: A Randomized Double Blind Clinical Trial Comparing Programed Intermittent Epidural Boluses (PIEB) Versus Patient Controlled Epidural Analgesia (PCEA) With Epidural or Combined Spinal-epidural (CSE) Technique
Brief Title: PIEB vs PCEA With Epidural or CSE Technique. A Randomized Double Blind Clinical Trial
Acronym: PIEB-CT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Emilia Guasch, Head of the Anesthesia and Intensive Care Department, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-004696-24
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Labor Epidural Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural analgesia (Experimental): Randomized allocation to receive patient controlled epidural analgesia or programed intermittent epidural boluses
  Interventions: Device: PCEA vs PIEB
- Epidural technique (Experimental): Randomized allocation to be punctioned a conventional epidural or a combined spinal-epidural technique
  Interventions: Procedure: Epidural vs CSE

INTERVENTIONS:
Device: PCEA vs PIEB — We evaluate the relation between the distribution of L-bupivacaine plus fentanyl in the epidural space and the incedence of breaktrough pain during labor
  Arms: Epidural analgesia
Procedure: Epidural vs CSE — We evaluate the relation between the type of epidural technique and the incedence of breaktrough pain during labor
  Arms: Epidural technique

SUMMARY:
The investigators have design a randomized double blind clinical trial to know the incidence of breaktrough pain (BP) in high-risk of BP parturients (nulliparous with early cervical dilation) comparing two epidural analgesic regimes: programed intermittent epidural boluses versus patient controlled epidural analgesia. The role of the epidural technique (epidural versus combined spinal-epidural) in the incidence of BP will be also evaluated.

DETAILED DESCRIPTION:
Women in labor receiving epidural analgesia may experience breakthrough pain (BP) that requires the use of additional medication and that is a source of dissatisfaction with the analgesic treatment for labor.

The investigators can define two types of BP: 'primary breakthrough pain' is the first moment when the patient requests analgesia during labor. 'Secondary breakthrough pain' can be defined as the time a previously effective epidural analgesia turns ineffective.

The BP may have multiple causes, such as delivery progression and catheter misplacement. There is no single pattern to provide adequate neuraxial analgesia for labor, but for certain patients and specific clinical situations some methods provide advantages over others.

The choice of a suitable system of epidural drug delivery has an important role in getting proper analgesia and a low incidence of breakthrough pain during labor. In order to develop preventive strategies for BP, some clinical scales to estimate its incidence rate have been described. Among risk factors for BP the investigators can include: Nulliparity, epidural catheter placement at an earlier cervical dilation, neonatal weight and technique performed (epidural versus combined spinal-epidural - CSE).

In addition, technological development has offered us new treatment modalities of pain management during childbirth have evolved recently to improve maternal satisfaction, as well as to treat and prevent BP: Patient Controlled Epidural Analgesia (PCEA) added or not to a continuous epidural infusion (CEI), computer integrated PCEA (CI-PCEA) and automatic or programed intermittent epidural boluses (PIEB).

Nowadays, there is no evidence about the best epidural analgesic treatment or the optimum epidural punction in order to reduce BP episodes and, hence, increase maternal satisfaction.

Therefore, the investigators have design a randomized double blind clinical trial to know the incidence of breaktrough pain (BP) in high-risk of BP parturients (nulliparous with early cervical dilation) comparing two epidural analgesic regimes added to a contiuous infusion of L-bupivacaine plus fentanyl: programed intermittent epidural boluses versus patient controlled epidural analgesia. The role of the epidural technique (epidural versus combined spinal-epidural) in the incidence of BP will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 40 years
2. Gestational age between 37 and 41 weeks
3. Singleton pregnancies
4. Nulliparity
5. Spontaneous or induced labor
6. Cervical dilation less than four centimeters

Exclusion Criteria:

1. Do not meet all the inclusion criteria
2. Do not consent to the study
3. Systemic medical pathologies as pre-eclampsia, insulin-treated gestational diabetes or multiple sclerosis that could influence medical decision during labour and/or make randomization unfeasible
4. Contraindication for neuraxial analgesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Incidence of breakthrough pain | Labor
  Evaluation of breakthough pain episodes since epidural punction to delivery

SECONDARY OUTCOMES:
Total epidural infusion volume | Labor
  Measurement of the total epidural infusion volume administered to the patient
Incidence of epidural failure | Labor
  Assesment the incidence of failed epdirual technique
Mode of delivery (spontaneous, intrumental and cesarean section) | Delivery
  Analysis of the potential relation of the interventions with the type of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Guasch, MD, PhD, Principal Investigator — Anesthesia and Intensive Care Department
Locations (1):
- University Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hess PE, Pratt SD, Lucas TP, Miller CG, Corbett T, Oriol N, Sarna MC. Predictors of breakthrough pain during labor epidural analgesia. Anesth Analg. 2001 Aug;93(2):414-8, 4th contents page. doi: 10.1097/00000539-200108000-00036. PMID 11473872
- [Background] Loubert C, Hinova A, Fernando R. Update on modern neuraxial analgesia in labour: a review of the literature of the last 5 years. Anaesthesia. 2011 Mar;66(3):191-212. doi: 10.1111/j.1365-2044.2010.06616.x. PMID 21320088
- [Background] van der Vyver M, Halpern S, Joseph G. Patient-controlled epidural analgesia versus continuous infusion for labour analgesia: a meta-analysis. Br J Anaesth. 2002 Sep;89(3):459-65. doi: 10.1093/bja/aef217. PMID 12402726
- [Background] American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Practice guidelines for obstetric anesthesia: an updated report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Anesthesiology. 2007 Apr;106(4):843-63. doi: 10.1097/01.anes.0000264744.63275.10. No abstract available. PMID 17413923
- [Background] Hogan Q. Distribution of solution in the epidural space: examination by cryomicrotome section. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):150-6. doi: 10.1053/rapm.2002.29748. PMID 11915061
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Halpern SH, Carvalho B. Patient-controlled epidural analgesia for labor. Anesth Analg. 2009 Mar;108(3):921-8. doi: 10.1213/ane.0b013e3181951a7f. PMID 19224805
- [Background] Stratmann G, Gambling DR, Moeller-Bertram T, Stackpole J, Pue AF, Berkowitz J. A randomized comparison of a five-minute versus fifteen-minute lockout interval for PCEA during labor. Int J Obstet Anesth. 2005 Jul;14(3):200-7. doi: 10.1016/j.ijoa.2004.12.008. PMID 15936187
- [Background] Sia AT, Lim Y, Ocampo CE. Computer-integrated patient-controlled epidural analgesia: a preliminary study on a novel approach of providing pain relief in labour. Singapore Med J. 2006 Nov;47(11):951-6. PMID 17075662
- [Background] Sng BL, Sia AT, Lim Y, Woo D, Ocampo C. Comparison of computer-integrated patient-controlled epidural analgesia and patient-controlled epidural analgesia with a basal infusion for labour and delivery. Anaesth Intensive Care. 2009 Jan;37(1):46-53. doi: 10.1177/0310057X0903700119. PMID 19157345
- [Background] Capogna G, Celleno D, Lyons G, Columb M, Fusco P. Minimum local analgesic concentration of extradural bupivacaine increases with progression of labour. Br J Anaesth. 1998 Jan;80(1):11-3. doi: 10.1093/bja/80.1.11. PMID 9505770
- [Background] Capogna G, Stirparo S. Techniques for the maintenance of epidural labor analgesia. Curr Opin Anaesthesiol. 2013 Jun;26(3):261-7. doi: 10.1097/ACO.0b013e328360b069. PMID 23563796
- [Background] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Background] Goodman SR, Smiley RM, Negron MA, Freedman PA, Landau R. A randomized trial of breakthrough pain during combined spinal-epidural versus epidural labor analgesia in parous women. Anesth Analg. 2009 Jan;108(1):246-51. doi: 10.1213/ane.0b013e31818f896f. PMID 19095858
- [Background] Boogmans T, Vertommen J, Valkenborgh T, Devroe S, Roofthooft E, Van de Velde M. Epidural neostigmine and clonidine improves the quality of combined spinal epidural analgesia in labour: a randomised, double-blind controlled trial. Eur J Anaesthesiol. 2014 Apr;31(4):190-6. doi: 10.1097/EJA.0b013e32836249e9. PMID 23959095